CLINICAL TRIAL: NCT03098381
Title: Alteration in Body Composition and Metabolic Profile Without Changes on Serum Leptin and Adiponectin Levels During Ramadan Fasting in Healthy Men
Brief Title: Alteration in Body Composition and Metabolic Profile During Ramadan Fasting in Healthy Men
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Suwimol Sapwarobol, Program Director, Nutrition and Dietetics Program, Chulalongkorn University
Other Study IDs: Nutrition and Dietetics Dept
Record Dates: First submitted 2017-03-15; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One of religious duties for all healthy adult Muslims is fasting during Ramadan, the ninth month of Islamic lunar calendar. In this month, Ramadan observance fasted (no food and drink) from dawn to dusk. Studies demonstrated daytime fasting may pose a positive significant effect on metabolic health. Thus, this present study aimed to determine the effect of Ramadan fasting on body composition, metabolic profile, serum leptin and adiponectin levels in healthy men.

DETAILED DESCRIPTION:
Outcome measurements were taken at before (baseline) and at the end of Ramadan (after Ramadan fasting) on body composition, metabolic profile (fasting plasma glucose, insulin, total cholesterol, HDL-c, LDL-c, triglycerides, and HOMA-IR), serum leptin and adiponectin, ratio of leptin to adiponectin in 27 healthy men (19-31 years) Muslim in Bangkok, Thailand.

Subjects Twenty-nine subjects fulfilled inclusion criteria including: age 19-40 years, Muslim men fasted completely, and no known of any metabolic-related diseases. Subjects with diseases and/or intake of any medication and dietary supplement, smoking, and alcohol drinking were excluded. After Ramadan fasting, 27 subjects completed the study.

The study protocol was approved by the Ethical Review Committee for Research Involving Human Research Participants, Health Science Group, Chulalongkorn University, Bangkok, Thailand (COA no. 136/2558).Written informed consent was obtained from all subjects prior to enrolling to the study. Subject's anonymity was preserved.

Study design Research visit was conducted at Faculty of Allied Health Sciences, Chulalongkorn University, Bangkok, Thailand at before (earlier days of Ramadan) and after (third week of Ramadan) to collect the outcome measurements including anthropometry, body composition, metabolic profile, serum leptin and adiponectin levels, and ratio of leptin to adiponectin. The dietary intake of 2 weekday and one weekend day and physical activity were recorded each week during Ramadan in food record booklet. Energy intake and macronutrients composition including carbohydrate, protein and fat will be analysed by registered dietitian.

Anthropometry and body composition measurements Weight, Body Mass Index (BMI), and percent body fat were measured at baseline (week-0) and the end of Ramadan fasting period (week-4). Body weight, and percent body fat mass were assessed using a constant current source with a high frequency current (50kHz, 500μA)-bioelectrical impedance analyzer (BIA) (MC-980MA body composition analyzer, TANITA corporation, Tokyo, JAPAN). The subject was requested to dress in light attire and bare feet. The 8 polar electrodes were positioned so that electric current was supplied from the electrodes on the tips of the toes of both feet and the fingertips of both hands, and voltage is measured on the heel of both feet and the near side of both hands. Body Mass Index (BMI) was calculated as weight/height2 (in kilograms per square meter). Waist and hip circumferences were measured by using a standard rounded tape at a point right above the iliac crest on the mid-axillary line at minimal respiration (for waist) and in a horizontal plane at the level of the maximal extension of the buttocks (for hip) to the nearest 1.0 cm.

Metabolic profile measurements Fasting blood samples were taken from vein puncture at before and after a period of Ramadan fasting. Separated serum samples were stored at - 80o C until analyses were performed. After withdrawal, blood samples were collected to determine the metabolic profile including plasma glucose, total cholesterol, high density lipoprotein-cholesterol (HDL-c), and triglycerides (TG) by enzymatic method while serum insulin levels were analyzed by Chemiluminescence. Low density lipoprotein-cholesterol (LDL-c) was estimated by using the Friedewald equation (LDL-c = [total cholesterol] - [HDL-c] - [TG]/5).22 Additionally, HOMA-IR was measured as fasting serum insulin (µIU/mL) x fasting plasma glucose (mmol/L)/22.5.23

Serum leptin and adiponectin measurements Serum leptin and adiponectin levels were assayed at the laboratory at Faculty of Allied Health Sciences, Chulalongkorn University. Serum leptin was measured using a commercially "Human Leptin Standard ABTS ELISA Development kit" (Peprotech, Inc., Rocky Hill, NJ, USA, Cat. no: 900-K90) at a wavelength of 405nm with correction set at 650nm, while serum adiponectin was measured using "Adiponectin (human) ELISA kit" (Enzo Life Sciences, Farmingdale, NY, USA, Cat. no: ALX-850-377) at a wavelength of 450nm with correction set at 630nm. Both serum leptin and adiponectin were measured by the enzyme-linked immunosorbent assay, and were carried out according to the manufacturer's procedure.

Statistical Analysis Data were expressed as frequency or percentage for descriptive; mean ± standard error mean (SEM), mean percentage change (% change) ± SEM for the continuous-normally distributed data; and median (range) for continuous-non normally distributed data. Paired student t-test, two related sample (Wilcoxon) test were employed for comparison of normally distributed and non-normally distributed data, respectively. Differences were considered as statistically significant for two-tailed of probability value or P less than 0.05. All analyses were performed using SPSS, version 16.0 (IBM, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* age 19-40 years
* Muslim men
* fasted completely during Ramadan
* no known of any metabolic-related diseases.

Exclusion Criteria:

* any diseases
* intake of any medication and dietary supplement
* smoking
* alcohol drinking

Ages: 19 Years to 40 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes
Study Population: 27 healthy men (19-31 years) Muslim
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
body composition | 1 months
  fat mass changes after 1 month of ramadan fasting in 27 participants

SECONDARY OUTCOMES:
Metabolic profile | 1 month
  cholesterol change after 1 month of ramadan fasting in 27 participants
Serum leptin and adiponectin measurements | 1 month
  concentrations of Leptin and Adiponectin changes after 1 month of ramadan fasting in 27 participants

CONTACTS AND LOCATIONS:
Overall Officials: Suwimol sapwarobol, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt J, Hotz HG, Foitzik T, Ryschich E, Buhr HJ, Warshaw AL, Herfarth C, Klar E. Intravenous contrast medium aggravates the impairment of pancreatic microcirculation in necrotizing pancreatitis in the rat. Ann Surg. 1995 Mar;221(3):257-64. doi: 10.1097/00000658-199503000-00007. PMID 7717779
- See also: Journal of human nutrition and dietetics — https://www.ncbi.nlm.nih.gov/labs/journals/j-hum-nutr-diet/